CLINICAL TRIAL: NCT03193307
Title: A Study to Investigate the Pharmacokinetic Drug-drug Interaction Following Oral Administration of Ethinylestradiol/Levonorgestrel (Microgynon®) and BI 409306 in Healthy Korean Premenopausal Female Subjects (an Open-label, Two-period, Fixed-sequence Study)
Brief Title: This Study Tests in Healthy Korean Women Which Effects BI 409306 and a Birth-control Pill Have on Each Other
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1289-0040
Record Dates: First submitted 2017-06-19; First posted 2017-06-20 (Actual); Results first posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-08

CONDITIONS: Healthy
MeSH Terms: interventions — BI 409306

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microgynon® 30 +BI 409306 then BI 409306 alone (Experimental): Run in period: Microgynon alone Treatment period: Microgynon® 30 +BI 409306 then BI 409306 alone
  Interventions: Drug: Microgynon® 30; Drug: BI 409306

INTERVENTIONS:
Drug: Microgynon® 30 — Run in period & Treatment Period
Drug: BI 409306 — Day 18 & 29 (Treatment Period)

SUMMARY:
The primary objective of this trial is to investigate the effect of multiple doses of ethinylestradiol / levonorgestrel (Microgynon®) on single dose pharmacokinetics of BI 409306 and the effect of single dose of BI 409306 on multiple dose pharmacokinetics of ethinylestradiol / levonorgestrel (Microgynon®)

ELIGIBILITY:
Inclusion Criteria:

* Healthy CYP2C19 PM genotyped premenopausal female subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests.
* Korean ethnicity according to the following criteria

  ;be a current Korean passport or national identification card holder, and have parents and grandparents who were all born in Korea
* Age of 19 to 40 years (incl.)
* Body Mass Index (BMI) of 18.5 to 25.0 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation
* Female subjects who meet any of the following criteria starting from at least 30 days before the first administration of trial medication and until 30 days after trial completion:

  * Use of adequate contraception, e.g. non-hormonal intrauterine device plus condom
  * Sexually abstinent
  * A vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
  * Surgically sterilised (including hysterectomy)

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minutes (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, oncologic or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial (including bioequivalence trial) where an investigational drug has been administered within 3 months prior to planned administration of trial medication
* Current smoker or ex-smoker who quit smoking less than 30 days prior to screening
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 20 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study.
* Any relevant finding of the gynaecological examination
* Thrombotic predisposition according to thrombophilic testing
* Existing or history of arterial thrombotic or embolic processes, conditions which predispose to them e.g. disorders of the clotting processes, valvular heart disease and atrial fibrillation
* Existing or history of confirmed venous thromboembolism, family history of venous thromboembolism, and other known risk factors for venous thromboembolism.
* Relevant varicosis
* Use of hormone-containing intrauterine device, depot injection or contraceptive implants
* Any history of relevant liver diseases (for instance, disturbances of liver function, jaundice or persistent itching during a previous pregnancy, Dubin-Johnson syndrome, Rotor syndrome, or previous or existing liver tumours)
* Any history of migraine with focal neurological symptoms

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open-label, two-period, fixed-sequence trial to investigate potential drug-drug interactions between BI 409306 and Microgynon® (ethinylestradiol and levonorgestrel). In run-in period, subjects were adjusted to Microgynon® treatment and in treatment period, BI 409306 and Microgynon® were either administered alone or in combination.
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects attended specialist sites which would then ensure that all subjects met all inclusion/exclusion criteria. Subjects were not to be entered to trial treatment if any one of the specific entry criteria were not met.
Groups:
- Microgynon® 30 + BI 409306 Then BI 409306 Alone: Participants were administered once daily orally one coated tablet (sugar coated) of Microgynon® 30 (containing 30 microgram (μg) ethinylestradiol (EE) and 150 μg levonorgestrel (LNG)) from Day 1 to Day 21.
  On Day 18 additionally to Microgynon®30, participants were also administered once daily orally one film coated tablet of 25 milligram (mg) of BI 409306 (Test 1 (T1)).
  On Day 29 participants were administered once daily orally one film coated tablet of 25 mg of BI 409306 (Reference 1 (R1)).
Period: Period 1 - Microgynon® 30 + BI 409306
Arm/Group | Microgynon® 30 + BI 409306 Then BI 409306 Alone
Started (Entered) | 16
Completed (Treated and completed) | 16
Not Completed | 0
Period: Period 2 - BI 409306 Alone
Arm/Group | Microgynon® 30 + BI 409306 Then BI 409306 Alone
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS) : The TS includes all subjects from the Entered set (ES; includes all entered subjects irrespective of treatment) who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Arm/Group | Microgynon® 30 + BI 409306 Then BI 409306 Alone
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: TS
  Years | 26.6 (4.43)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: TS
  Participants
    Female | 16
    Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: TS
  Participants
    American Indian or Alaska Native | 0
    Asian | 16
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 409306 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: AUC0-tz , area under the concentration-time curve of BI 409306 in plasma over the time interval from 0 to the last quantifiable concentration is presented.
  Geometric Least Squares Mean and adjusted geometric standard error were derived from an Analysis of variance (ANOVA) model which included random effect for 'subject' and fixed effect for 'treatment'.
  Pharmacokinetics samples were collected 10 minutes (min) pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 14, 24, 36, 48 and 72 hours (h) after single oral administration of 1 tablet of 25 mg BI 409306 together with 1 tablet of Microgynon® 30 (Day 18) and after single administration of one tablet of 25 mg BI 409306 alone (Day 29).
Time Frame: PK samples were collected 10 min pre-dose and up to 72 h after administration of BI 409306 together with Microgynon® 30 (Day 18) and up to 72 h after administration of BI 409306 alone (Day 29).
Population: Pharmacokinetic (PK) set (PKS): The PKS included all subjects in the treated set (TS) who provided at least one primary or secondary PK parameter value for one period to the statistical assessment and was not excluded from the study as predefined in the Trial statistical analysis plan (TSAP).
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomoles*hour/Litre [nmol*h/L]
Groups:
- BI 409306 + Microgynon® 30 (T1): Subjects were administered orally 1 tablet of 25 milligram (mg) BI 409306 together with 1 tablet Microgynon® 30 on Day 18 (Test 1 (T1)).
- BI 409306 Alone (R1): Subjects were administered orally 1 tablet of 25 mg BI 409306 alone on Day 29 (Reference 1 (R1)).
Arm/Group | BI 409306 + Microgynon® 30 (T1) | BI 409306 Alone (R1)
Number analyzed (Participants) | 16 | 16
nanomoles*hour/Litre [nmol*h/L] | 5931.13 (NA) — Adjusted geometric standard error=1.084. | 3871.50 (NA) — Adjusted geometric standard error=1.084.
Statistical Analysis 1: Comparison: BI 409306 + Microgynon® 30 (T1) vs BI 409306 Alone (R1); Test type: Other; Geometric Mean (T1/R1) ratio (%) = 153.20, 90% CI 2-sided [134.34 to 174.70] — Analysis of variance (ANOVA) model including random effect for 'subject' and fixed effect for 'treatment' was used. Intra-individual geometric coefficient of variation (gCV [%]) =21.4

2. Primary Outcome: Maximum Measured Concentration of BI 409306 in Plasma (Cmax)
Description: Cmax, maximum measured concentration of BI 409306 in plasma is presented. Geometric Least Squares Mean and adjusted geometric standard error were derived from an Analysis of variance (ANOVA) model which included random effect for 'subject' and fixed effect for 'treatment'.
  Pharmacokinetics samples were collected 10 minutes (min) pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 14, 24, 36, 48 and 72 hours (h) after single oral administration of 1 tablet of 25 mg BI 409306 together with 1 tablet of Microgynon® 30 (Day 18) and after single administration of one tablet of 25 mg BI 409306 alone (Day 29).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomoles/Litre [nmol/L]
Arm/Group | BI 409306 + Microgynon® 30 (T1) | BI 409306 Alone (R1)
Number analyzed (Participants) | 16 | 16
nanomoles/Litre [nmol/L] | 1786.026 (NA) — Adjusted geometric standard error=1.054. | 1540.816 (NA) — Adjusted geometric standard error=1.054.
Statistical Analysis 1: Comparison: BI 409306 + Microgynon® 30 (T1) vs BI 409306 Alone (R1); Test type: Other; Geometric Mean (T1/R1) ratio (%) = 115.91, 90% CI 2-sided [104.559 to 128.502] — Analysis of variance (ANOVA) including random effect for 'subject' and fixed effect for 'treatment' was used. Intra-individual geometric coefficient of variation (gCV [%]) = 16.7

3. Primary Outcome: Area Under the Concentration-time Curve of Ethinylestradiol in Plasma Over the Time Interval From 0 to 24 Hour at Steady State (AUC0-24,ss)
Description: AUC0-24,ss, area under the concentration-time curve of the ethinylestradiol in plasma over the time interval from 0 to 24 hour at steady state.
  Geometric Least Squares Mean and adjusted geometric standard error were derived from an Analysis of variance (ANOVA) model which included random effect for 'subject' and fixed effect for 'treatment'.
  Pharmacokinetics samples were collected 10 minutes (min) pre-dose, 0.5, 1, 1.5, 2, 4, 8, 14 and 24 hours (h) after single oral administration of 1 tablet Microgynon® 30 (Day 17) and after single administration of 1 tablet Microgynon® 30 together with one tablet of 25 mg BI 409306 (Day 18).
Time Frame: PK samples were collected 10 min pre-dose and up to 24 h after administration of Microgynon® 30 (Day 17) and up to 24 h after administration of Microgynon® 30 together with BI 409306 (Day 18).
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: Picograms*hour/millilitre [pg*h/mL]
Groups:
- Microgynon® 30 + BI 409306 (T2): Subjects were administered orally 1 tablet of Microgynon® 30 (at steady state) together with 1 tablet of 25 mg BI 409306 on Day 18 (Test 2 (T2)).
- Microgynon® 30 Alone (R2): Subjects were administered orally 1 tablet of Microgynon® 30 alone on Day 17 (at steady state) (Reference 2 (R2)).
Arm/Group | Microgynon® 30 + BI 409306 (T2) | Microgynon® 30 Alone (R2)
Number analyzed (Participants) | 16 | 16
Picograms*hour/millilitre [pg*h/mL] | 921.880 (NA) — Adjusted geometric standard error=1.104. | 879.521 (NA) — Adjusted geometric standard error=1.104.
Statistical Analysis 1: Comparison: Microgynon® 30 + BI 409306 (T2) vs Microgynon® 30 Alone (R2); Test type: Other; Geometric Mean (T2/R2) ratio (%) = 104.82, 90% CI 2-sided [102.092 to 107.613] — Analysis of variance (ANOVA) model including random effect for 'subject' and fixed effect for 'treatment' was used. Intra-individual geometric coefficient of variation (gCV [%]) =4.3

4. Primary Outcome: Area Under the Concentration-time Curve of Levonorgestrel in Plasma Over the Time Interval From 0 to 24 Hour at Steady State (AUC0-24,ss)
Description: AUC0-24,ss, area under the concentration-time curve of the levonorgestrel in plasma over the time interval from 0 to 24 hour at steady state.
  Geometric Least Squares Mean and adjusted geometric standard error were derived from an Analysis of variance (ANOVA) model which included random effect for 'subject' and fixed effect for 'treatment'.
  Pharmacokinetics samples were collected 10 minutes (min) pre-dose, 0.5, 1, 1.5, 2, 4, 8, 14 and 24 hours (h) after single oral administration of 1 tablet Microgynon® 30 (Day 17) and after single administration of 1 tablet Microgynon® 30 together with one tablet of 25 mg BI 409306 (Day 18).
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: Picograms*hour/millilitre [pg*h/mL]
Arm/Group | Microgynon® 30 + BI 409306 (T2) | Microgynon® 30 Alone (R2)
Number analyzed (Participants) | 16 | 16
Picograms*hour/millilitre [pg*h/mL] | 86110.14 (NA) — Adjusted geometric standard error=1.108. | 83791.03 (NA) — Adjusted geometric standard error=1.108.
Statistical Analysis 1: Comparison: Microgynon® 30 + BI 409306 (T2) vs Microgynon® 30 Alone (R2); Test type: Other; Geometric Mean (T2/R2) ratio (%) = 102.77, 90% CI 2-sided [100.66 to 104.92] — Analysis of variance (ANOVA) model including random effect for 'subject' and fixed effect for 'treatment' was used. Intra-individual geometric coefficient of variation (gCV [%]) = 3.3

5. Primary Outcome: Maximum Measured Concentration of Ethinylestradiol in Plasma at Steady State (Cmax,ss)
Description: Cmax,ss, maximum measured concentration of ethinylestradiol in plasma at steady state is presented.
  Geometric Least Squares Mean and adjusted geometric standard error were derived from an Analysis of variance (ANOVA) model which included random effect for 'subject' and fixed effect for 'treatment'.
  Pharmacokinetics samples were collected 10 minutes (min) pre-dose, 0.5, 1, 1.5, 2, 4, 8, 14 and 24 hours (h) after single oral administration of 1 tablet Microgynon® 30 (Day 17) and after single administration of 1 tablet Microgynon® 30 together with one tablet of 25 mg BI409306 (Day 18).
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: Picograms/millilitre [pg/mL]
Arm/Group | Microgynon® 30 + BI 409306 (T2) | Microgynon® 30 Alone (R2)
Number analyzed (Participants) | 16 | 16
Picograms/millilitre [pg/mL] | 112.405 (NA) — Standard error is actually adjusted geometric standard error. Adjusted geometric standard error=1.089. | 98.500 (NA) — Standard error is actually adjusted geometric standard error. Adjusted geometric standard error=1.089.
Statistical Analysis 1: Comparison: Microgynon® 30 + BI 409306 (T2) vs Microgynon® 30 Alone (R2); Test type: Other; Geometric Mean (T2/R2) ratio (%) = 114.12, 90% CI 2-sided [109.266 to 119.183] — Analysis of variance (ANOVA) model including random effect for 'subject' and fixed effect for 'treatment' was used. Intra-individual geometric coefficient of variation (gCV [%])=7.0

6. Primary Outcome: Maximum Measured Concentration of Levonorgestrel in Plasma at Steady State (Cmax,ss)
Description: Cmax,ss, maximum measured concentration of levonorgestrel in plasma at steady state is presented.
  Geometric Least Squares Mean and adjusted geometric standard error were derived from an Analysis of variance (ANOVA) model which included random effect for 'subject' and fixed effect for 'treatment'.
  Pharmacokinetics samples were collected 10 minutes (min) pre-dose, 0.5, 1, 1.5, 2, 4, 8, 14 and 24 hours (h) after single oral administration of 1 tablet Microgynon® 30 (Day 17) and after single administration of 1 tablet Microgynon® 30 together with one tablet of 25 mg BI409306 (Day 18).
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: Picograms/millilitre [pg/mL]
Arm/Group | Microgynon® 30 + BI 409306 (T2) | Microgynon® 30 Alone (R2)
Number analyzed (Participants) | 16 | 16
Picograms/millilitre [pg/mL] | 7867.89 (NA) — Adjusted geometric standard error=1.084. | 7107.42 (NA) — Adjusted geometric standard error=1.084.
Statistical Analysis 1: Comparison: Microgynon® 30 + BI 409306 (T2) vs Microgynon® 30 Alone (R2); Test type: Other; Geometric Mean (T2/R2) ratio (%) = 110.70, 90% CI 2-sided [105.80 to 115.83] — Analysis of variance (ANOVA) model including random effect for 'subject' and fixed effect for 'treatment' was used. Intra-individual geometric coefficient of variation (gCV [%]) = 7.3

7. Secondary Outcome: Area Under the Concentration-time Curve of BI 409306 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-infinity)
Description: AUC0-infinity, area under the concentration-time curve of BI 409306 in plasma over the time interval from 0 extrapolated to infinity is presented.
  Geometric Least Squares Mean and adjusted geometric standard error were derived from an Analysis of variance (ANOVA) model which included random effect for 'subject' and fixed effect for 'treatment'.
  Pharmacokinetics samples were collected 10 minutes (min) pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 14, 24, 36, 48 and 72 hours (h) after single oral administration of 1 tablet of 25 mg BI 409306 together with 1 tablet of Microgynon® 30 (Day 18) and after single administration of 1 tablet of 25 mg BI 409306 alone (Day 29).
Time Frame: PK samples were collected 10 min pre-dose and up to 72h after administration of BI 409306 together with Microgynon® 30 (Day 18) and up to 72 h after administration of BI 409306 alone (Day 29).
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: Nanomole*hour/milllilitre [nmol*h/mL]
Arm/Group | BI 409306 + Microgynon® 30 (T1) | BI 409306 Alone (R1)
Number analyzed (Participants) | 15 | 16
Nanomole*hour/milllilitre [nmol*h/mL] | 6000.32 (NA) — Adjusted geometric standard error=1.086. | 3892.47 (NA) — Adjusted geometric standard error=1.086.
Statistical Analysis 1: Comparison: BI 409306 + Microgynon® 30 (T1) vs BI 409306 Alone (R1); Test type: Other; Geometric Mean (T1/R1) ratio (%) = 154.15, 90% CI 2-sided [133.81 to 177.58] — Analysis of variance (ANOVA) model including random effect for 'subject' and fixed effect for 'treatment' was used. Intra-individual geometric coefficient of variation (gCV [%]) = 22.4

ADVERSE EVENTS:
Time Frame: From first drug administration until 6 days after last drug administration, up to 35 days.
Description: This subject set included all subjects from the entered set (all entered subjects, whether treated or not) who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Groups:
- Total BI409306: Subjects were administered orally 1 tablet of 25 mg BI 409306 alone on Day 29 or 1 tablet of 25 mg BI 409306 together with 1 tablet Microgynon® 30 on Day 18.
Arm/Group | Microgynon® 30 Alone (R2) | BI 409306 + Microgynon® 30 (T1) | BI 409306 Alone (R1) | Total BI409306 | Microgynon® 30 + BI 409306 Then BI 409306 Alone
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 9/16 | 11/16 | 12/16 | 14/16 | 15/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Microgynon® 30 Alone (R2) (N=16) | BI 409306 + Microgynon® 30 (T1) (N=16) | BI 409306 Alone (R1) (N=16) | Total BI409306 (N=16) | Microgynon® 30 + BI 409306 Then BI 409306 Alone (N=16)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 1
Visual brightness (Eye disorders) | 0 | 7 | 10 | 10 | 10
Abnormal sensation in eye (Eye disorders) | 0 | 1 | 0 | 1 | 1
Conjunctival hyperaemia (Eye disorders) | 0 | 1 | 0 | 1 | 1
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 1 | 1
Photopsia (Eye disorders) | 0 | 1 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 2 | 4 | 4
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Catheter site pain (General disorders) | 0 | 1 | 0 | 1 | 1
Feeling cold (General disorders) | 0 | 1 | 0 | 1 | 1
Vessel puncture site erythema (General disorders) | 0 | 1 | 0 | 1 | 1
Tooth injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 2 | 3 | 5 | 5
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 3 | 3
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2 | 2
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT03193307/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT03193307/SAP_001.pdf